CLINICAL TRIAL: NCT00002191
Title: A Double-Blind, Placebo-Controlled Trial of Albendazole in HIV-Positive Patients With Intestinal Microsporidiosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SmithKline Beecham (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 274A; SK 62979/029; GHBA 659
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-07

CONDITIONS: Protozoan Infections; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Placebos; Protozoan Infections; Intestinal Diseases; Albendazole; Microsporida; Anthelmintics
MeSH Terms: conditions — Protozoan Infections; HIV Infections; AIDS-Related Opportunistic Infections; Intestinal Diseases | interventions — Albendazole

INTERVENTIONS:
Drug: Albendazole

SUMMARY:
To evaluate the efficacy (stool frequency) and safety (adverse experiences) of albendazole, administered for 28 days, compared to placebo and for 62 days in open-label fashion, in treating intestinal microsporidiosis in HIV-positive patients. To assess the effect of albendazole on stool volume, weight gain, microsporidial counts in small bowel biopsies, and on the relationship between microsporidial counts in stool and stool frequency and volume. To correlate microsporidial counts with the clinical course of microsporidiosis.

DETAILED DESCRIPTION:
In the double-blind portion of study, patients receive albendazole or placebo for 28 days; in the open-label portion of study, patients receive albendazole for 62 days.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* If coincident enteric pathogens that are not eradicable (i.e., Mycobacterium avium complex) are detected, they should be treated appropriately and the patient must be on a stable regimen of therapy for at least two weeks.

Allowed:

* Patients taking antidiarrheal medications must be on a stable regimen for at least seven days prior to randomization.
* Patients taking other concomitant medications, including antiretrovirals, must be on a stable regimen for two weeks prior to randomization.

Patients must have:

* HIV positive status. Written documentation (for example, patient's chart) of HIV diagnosis is acceptable in lieu of repeat testing. Confirmation by Western blot is not necessary.
* Biopsy-proven microsporidiosis of the fourth portion of the duodenum or proximal jejunum within 90 days before randomization.
* Average of > 3 liquid bowel movements per day over 7 consecutive days immediately prior to randomization, with an average volume > 500 ml per day over three or more consecutive days immediately prior to randomization, as documented by data collected in a daily diary. NOTE:
* Patients receiving antidiarrheal therapy must meet these criteria despite such therapy.
* History of an average of > 3 liquid bowel movements per day for three additional weeks immediately preceding the 7-day period described above (for a total of four weeks), as documented in the patient's chart.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Grade 4 neutropenia.
* Decompensated liver disease.
* Positive toxin analysis for C. difficile.
* Positive microscopic examination for Giardia lamblia, Entamoeba histolytica, and Isospora belli.
* Positive on culture for Shigella, Salmonella, Yersinia and Campylobacter.
* Positive fluorescent antibody test for Cryptosporidium.
* Evidence of CMV on small bowel biopsy, flexible sigmoidoscopic or colonoscopic biopsies within 90 days of randomization.
* Any other condition that, in the opinion of the investigator, makes the patient unsuitable for study entry.

Patients with the following prior conditions are excluded:

Hypersensitivity to albendazole.

Prior Medication:

Excluded:

* Use of potential antiprotozoal drugs, e.g., mebendazole or metronidazole, within one week prior to enrollment.
* Receipt of albendazole during the one month prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - San Francisco Gen Hosp / Div of GI, San Francisco, California
  - Davies Med Ctr, San Francisco, California
  - George Washington Univ 5-403A, Washington D.C., District of Columbia
  - Deaconess Hosp / Harvard Med School / Infect Disease, Boston, Massachusetts
  - New York Univ, New York, New York
  - Saint Luke's Hosp / Services and Research 1301, New York, New York